CLINICAL TRIAL: NCT04987398
Title: Analysis of Ventilation Weaning Strategies and Correlation to Outcomes in Tracheostomized Patients in the Intensive Care Unit of the Lausanne University Hospital
Brief Title: Ventilation Weaning Strategies and Correlation to Outcomes in Tracheostomized Patients in the Lausanne ICU
Status: Completed | Type: Observational
Sponsor: Piquilloud Imboden Lise (Other)
Responsible Party: Sponsor-Investigator, Piquilloud Imboden Lise, Sponsor-Investigator, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Other Study IDs: TRACH-CHANGE
Record Dates: First submitted 2021-07-12; First posted 2021-08-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Failure; Tracheostomy Complication
Keywords: Tracheostomy; Ventilation weaning; spontaneous breathing trial
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intubation for respiratory reasons: All patients who were intubated for respiratory reasons (i.e. acute respiratory distress syndrome, pneumonias, pleural effusions for example)
- Intubation for neurological reasons: All patients who were intubated for neurological reasons (i.e. stroke, intracranial bleeding, cervical fracture with tetraparesia for example)
- Intubation for other reasons: All patients who were intubated for other reasons than respiratory or neurological (i.e. intubation before surgery, cardiac arrest, hemodynamic instability and polytraumatism without respiratory distress or neurological pathology necessitating intubation)

SUMMARY:
This retrospective study aims to study characteristics of patients tracheotomized in the Lausanne ICU, both overall and by primary reasons of intubation. Ventilation data both before and after tracheotomy, weaning technique and timing are studied in this retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized in the Lausanne ICU between May 1st 2017 and November 31st 2018 with a tracheotomy and mechanically ventilated more than 72 hours.

Exclusion Criteria:

* Presence of a know opposition to participation to research projects
* Patient tracheostomized specifically for ENT (ear-nose-throat) reason
* Burn victim
* Patient tracheostomized before his/her admission to the Lausanne ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Lausanne ICU between May1st and November 31st who had a tracheotomy and were ventilated for more than 72 hours were screened for exclusion criterias. 147 patients were screened and 80 patients were included.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Time from intubation to tracheotomy | Once, between time of intubation to time of tracheotomy, up to 60 days
  Calculated from clinical information system (time of intubation, time of tracheotomy), calculated in hours

SECONDARY OUTCOMES:
Age | At ICU admission
  Collected from electronic patient files.
Weight | At ICU admission
  Collected from electronic patient files.
Height | At ICU admission
  Collected from electronic patient files.
Body mass index | At ICU admission
  Calculated from weight and height
Predicted body weight (PBW) | At ICU admission
  Calculated as such :
  Adult male: 50 + 0.91 (Height cm -152.4) / Adult female: 45 + 0.91 (Height cm -152.4)
SOFA score (admission) | At ICU admission
  Calculated at admission
Clinical Frailty Score | At ICU admission
  Calculated at ICU admission
Charlson comorbidity index | At ICU admission
  Calculated at ICU admission
Comorbidities | At ICU admission
  Collected at ICU admission
Ventilation modalities and settings from intubation to tracheotomy | Once every day at 8am, between day after intubation to day before tracheotomy, up to 60 days
  Ventilation modalities and settings recolted from electronic patient files.
Sedation opioid use from intubation to tracheotomy | Once every day at 8am and at time of minimal and maximal value, between day of intubation to day of tracheotomy, up to 60 days
  Sedation use collected from electronic patient files.
Opioid use from intubation to tracheotomy | Once every day at 8am and at time of minimal and maximal value, between day of intubation to day of tracheotomy, up to 60 days
  Opioid use collected from electronic patient files.
Neuromuscular blocking agent use from intubation to tracheotomy | Once every day at 8am and at time of minimal and maximal value, between day of intubation to day of tracheotomy, up to 60 days
  Neuromuscular blocking agent use collected from electronic patient files.
Tracheotomy time | At time of tracheotomy, once, up to 60 days after intubation day
  Collected from electronic patient files (day and hour)
Tracheotomy type (percutaneous, surgical) | At time of tracheotomy, once, up to 60 days after intubation day
  Collected from electronic patient files.
Ventilation settings and modalities from day of tracheotomy | 2 hours before tracheotomy
  Collected from electronic patient files.
SOFA score (tracheotomy day) | Once, on the day of tracheotomy (worst value of the day of tracheotomy), up to 60 days after intubation day
  Calculated from electronic patient files.
Ventilation modalities and settings from tracheotomy to mechanical ventilation weaning | Once per day, from day of tracheotomy to mechanical ventilation weaning, up to 60 days
  Ventilation modalities and settings collected from electronic patient files.
Tracheotomy weaning strategies from tracheotomy to mechanical ventilation weaning | Once every day at 8am and at time of minimal and maximal value, from day of tracheotomy to day of mechanical ventilation weaning, up to 31 days
  Data collected from electronic patient files.
Physical therapy sessions from tracheotomy to mechanical ventilation weaning | Once every day at 8am and at time of minimal and maximal value, from day of tracheotomy to day of mechanical ventilation weaning, up to 31 days
  Data collected from electronic patient files.
Mechanical ventilation weaning day | Once (day 3 in a row of less than 12 hours of mechanical ventilation), up to 31 days after tracheotomy day
  Data collected from electronic patient files.
SOFA score (mechanical ventilation weaning day) | Once (3rd consecutive day with less than 12-h of mechanical ventilation), up to 31 days after tracheotomy day
  Calcutated from electronic patient files.
Ventilation modalities and settings from mechanical ventilation weaning day to decannulation or ICU discharge or death | Once every day at 8am and at time of minimal and maximal value, from day of mechanical ventilation weaning to decannulation or ICU discharge or death, up to 31 days
  Collected from electronic patient files.
Physical therapy sessions from mechanical ventilation weaning day to decannulation or ICU discharge or death | Once every day at 8am and at time of minimal and maximal value, from day of mechanical ventilation weaning to decannulation or ICU discharge or death, up to 31 days
  Collected from electronic patient files.
Hospital stay duration | Once, between day of hospital admission to day of hospital discharge, up to 2 years
  Collected from electronic patient files and discharge letters
Outcome and specific treatments in ICU | Once, between day of hospital admission to day of hospital discharge, up to 2 years
  Data recolted from electronic patient files
Correlation of ventilation settings and modalities and tracheotomy weaning strategies | Once, between day of hospital admission to day of hospital discharge, up to 2 years
  Collected from electronic patient files and discharge letters

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andriolo BN, Andriolo RB, Saconato H, Atallah AN, Valente O. Early versus late tracheostomy for critically ill patients. Cochrane Database Syst Rev. 2015 Jan 12;1(1):CD007271. doi: 10.1002/14651858.CD007271.pub3. PMID 25581416
- [Background] Arabi Y, Haddad S, Shirawi N, Al Shimemeri A. Early tracheostomy in intensive care trauma patients improves resource utilization: a cohort study and literature review. Crit Care. 2004 Oct;8(5):R347-52. doi: 10.1186/cc2924. Epub 2004 Aug 23. PMID 15469579
- [Background] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Background] Burns KEA, Soliman I, Adhikari NKJ, Zwein A, Wong JTY, Gomez-Builes C, Pellegrini JA, Chen L, Rittayamai N, Sklar M, Brochard LJ, Friedrich JO. Trials directly comparing alternative spontaneous breathing trial techniques: a systematic review and meta-analysis. Crit Care. 2017 Jun 1;21(1):127. doi: 10.1186/s13054-017-1698-x. PMID 28576127
- [Background] Delaney A, Bagshaw SM, Nalos M. Percutaneous dilatational tracheostomy versus surgical tracheostomy in critically ill patients: a systematic review and meta-analysis. Crit Care. 2006;10(2):R55. doi: 10.1186/cc4887. PMID 16606435
- [Background] McCredie VA, Alali AS, Scales DC, Adhikari NK, Rubenfeld GD, Cuthbertson BH, Nathens AB. Effect of Early Versus Late Tracheostomy or Prolonged Intubation in Critically Ill Patients with Acute Brain Injury: A Systematic Review and Meta-Analysis. Neurocrit Care. 2017 Feb;26(1):14-25. doi: 10.1007/s12028-016-0297-z. PMID 27601069
- [Background] Mehta AB, Walkey AJ, Curran-Everett D, Douglas IS. One-Year Outcomes Following Tracheostomy for Acute Respiratory Failure. Crit Care Med. 2019 Nov;47(11):1572-1581. doi: 10.1097/CCM.0000000000003959. PMID 31397716
- [Background] Young D, Harrison DA, Cuthbertson BH, Rowan K; TracMan Collaborators. Effect of early vs late tracheostomy placement on survival in patients receiving mechanical ventilation: the TracMan randomized trial. JAMA. 2013 May 22;309(20):2121-9. doi: 10.1001/jama.2013.5154. PMID 23695482